CLINICAL TRIAL: NCT06515860
Title: Observational Trial of Liquid Biopsy for Malignant Peripheral Nerve Sheath Tumor (MPNST) Among Participants With Neurofibromatosis Type 1
Brief Title: Neurofibromatosis Type 1 Tumor Early Detection Study
Acronym: NF1-TED
Status: Recruiting | Type: Observational
Sponsor: David Miller (Other)
Responsible Party: Sponsor-Investigator, David Miller, Principal Investigator, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Other Study IDs: 23-380; 23-380 (Other: Dana Farber/Harvard Cancer Center IRB)
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromatosis Type 1; Neurofibromatosis 1; Plexiform Neurofibroma; Plexiform Neurofibromas; Malignant Peripheral Nerve Sheath Tumor; Malignant Peripheral Nerve Sheath Tumors; Atypical Neurofibroma
Keywords: Liquid biopsy; Cancer surveillance; Tumor early detection
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Neurofibrosarcoma | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh blood will be processed at receipt into blood products (e.g., plasma) or frozen whole. Plasma aliquots and frozen whole blood will be stored in a -80°C or -20°C freezer until distribution. Frozen tissue will be received, weighed, and banked in a liquid nitrogen vapor phase freezer. At the end of the study, selected blood and tissue samples may be pulled for nucleic acid extraction. Prior to extracting nucleic acid from tissue, a pathology quality control review will determine the %tumor and %necrotic tumor, as well as confirm concordance with the institutional diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Liquid biopsy for MPNST development — Participants will be asked to complete a blood sample (liquid biopsy) at baseline (15 mL, approximately 1 tablespoon) and every 6 months (10 mL) for the five-year follow-up period.

SUMMARY:
The goal of this observational study is to determine if a liquid biopsy (i.e. blood test) is an effective clinical tool for monitoring the development of malignant peripheral nerve sheath tumor (MPNST) among adults (18 years and older) with Neurofibromatosis Type 1 (NF1), compared to the current standard of care. The main questions it aims to answer are:

How effective is liquid biopsy compared to the current standard of care (clinical surveillance and imaging) for early detection of MPNST development among people with NF1? Can liquid biopsy offer a cost-effective method for early detection of MPNST in people with NF1? Also, can liquid biopsy provide earlier detection that potentially leads to better outcomes? Also, can offering liquid biopsy improve access to care for people experiencing barriers to access (such as minority populations or people in rural areas)?

At baseline, participants will be asked to:

* Complete surveys to provide their demographic and NF1-related health information.
* Report whether or not they are experiencing MPNST-related symptoms.
* Provide blood samples (15 mL blood total between three tubes, which is approximately one tablespoon).

Every six months during the five-year follow-up period, participants will be asked to:

* Complete additional surveys to report whether or not they are experiencing MPNST-related symptoms and/or if they have been diagnosed with a new MPNST.
* Provide an additional blood sample (10 mL blood total in one tube).

If diagnosed with an MPNST by their healthcare provider during the follow-up period, participants will be asked to:

* Complete an additional survey regarding their diagnosis and symptoms.
* Provide an additional blood sample (10 mL blood in one tube).
* In parallel, the study team will request a sample of tumor tissue from the care provider, if available.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older (adults only)
* Neurofibromatosis Type 1 (NF1) diagnosis (2021 Revised Diagnostic Criteria, PMID: 34012067)
* History of plexiform neurofibroma (PN)
* Able to read and understand English or Spanish
* Live in the USA

Exclusion Criteria:

* Are children (younger than 18 years old)
* Do not have NF1
* Have no evidence of PN
* Are not able to read and understand English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults with NF1 who live in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Timing of MPNST detection by liquid biopsy | From enrollment to the end of the five-year follow-up period
  Comparison will be made between date of clinical diagnosis versus the date when the tumor could be detected in a liquid biopsy sample.

SECONDARY OUTCOMES:
Number of participants with new MPNST | From enrollment to the end of the five-year follow-up period
  New MPNST diagnosed by healthcare provider (Yes/No). The number of participants who develop an MPNST will be compared to the overall size of the cohort.

CONTACTS AND LOCATIONS:
Overall Officials: David T Miller, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Investigators conducting the analysis at the end of the follow-up period will need access to IPD, but the plan to share IPD is not yet written.

REFERENCES:
- [Background] Miettinen MM, Antonescu CR, Fletcher CDM, Kim A, Lazar AJ, Quezado MM, Reilly KM, Stemmer-Rachamimov A, Stewart DR, Viskochil D, Widemann B, Perry A. Histopathologic evaluation of atypical neurofibromatous tumors and their transformation into malignant peripheral nerve sheath tumor in patients with neurofibromatosis 1-a consensus overview. Hum Pathol. 2017 Sep;67:1-10. doi: 10.1016/j.humpath.2017.05.010. Epub 2017 May 24. PMID 28551330
- [Background] Klein EA, Richards D, Cohn A, Tummala M, Lapham R, Cosgrove D, Chung G, Clement J, Gao J, Hunkapiller N, Jamshidi A, Kurtzman KN, Seiden MV, Swanton C, Liu MC. Clinical validation of a targeted methylation-based multi-cancer early detection test using an independent validation set. Ann Oncol. 2021 Sep;32(9):1167-1177. doi: 10.1016/j.annonc.2021.05.806. Epub 2021 Jun 24. PMID 34176681
- [Background] Chaudhuri AA, Chabon JJ, Lovejoy AF, Newman AM, Stehr H, Azad TD, Khodadoust MS, Esfahani MS, Liu CL, Zhou L, Scherer F, Kurtz DM, Say C, Carter JN, Merriott DJ, Dudley JC, Binkley MS, Modlin L, Padda SK, Gensheimer MF, West RB, Shrager JB, Neal JW, Wakelee HA, Loo BW Jr, Alizadeh AA, Diehn M. Early Detection of Molecular Residual Disease in Localized Lung Cancer by Circulating Tumor DNA Profiling. Cancer Discov. 2017 Dec;7(12):1394-1403. doi: 10.1158/2159-8290.CD-17-0716. Epub 2017 Sep 24. PMID 28899864
- [Background] Pemov A, Li H, Presley W, Wallace MR, Miller DT. Genetics of human malignant peripheral nerve sheath tumors. Neurooncol Adv. 2019 Nov 28;2(Suppl 1):i50-i61. doi: 10.1093/noajnl/vdz049. eCollection 2020 Jul. PMID 32642732
- [Background] Cortes-Ciriano I, Steele CD, Piculell K, Al-Ibraheemi A, Eulo V, Bui MM, Chatzipli A, Dickson BC, Borcherding DC, Feber A, Galor A, Hart J, Jones KB, Jordan JT, Kim RH, Lindsay D, Miller C, Nishida Y, Proszek PZ, Serrano J, Sundby RT, Szymanski JJ, Ullrich NJ, Viskochil D, Wang X, Snuderl M, Park PJ, Flanagan AM, Hirbe AC, Pillay N, Miller DT; Genomics of MPNST (GeM) Consortium. Genomic Patterns of Malignant Peripheral Nerve Sheath Tumor (MPNST) Evolution Correlate with Clinical Outcome and Are Detectable in Cell-Free DNA. Cancer Discov. 2023 Mar 1;13(3):654-671. doi: 10.1158/2159-8290.CD-22-0786. PMID 36598417
- [Background] Mautner VF, Asuagbor FA, Dombi E, Funsterer C, Kluwe L, Wenzel R, Widemann BC, Friedman JM. Assessment of benign tumor burden by whole-body MRI in patients with neurofibromatosis 1. Neuro Oncol. 2008 Aug;10(4):593-8. doi: 10.1215/15228517-2008-011. Epub 2008 Jun 17. PMID 18559970
- [Background] Pemov A, Li H, Patidar R, Hansen NF, Sindiri S, Hartley SW, Wei JS, Elkahloun A, Chandrasekharappa SC; NISC Comparative Sequencing Program; Boland JF, Bass S; NCI DCEG Cancer Genomics Research Laboratory; Mullikin JC, Khan J, Widemann BC, Wallace MR, Stewart DR. The primacy of NF1 loss as the driver of tumorigenesis in neurofibromatosis type 1-associated plexiform neurofibromas. Oncogene. 2017 Jun 1;36(22):3168-3177. doi: 10.1038/onc.2016.464. Epub 2017 Jan 9. PMID 28068329
- See also: Neurofibromatosis Type 1 Tumor Early Detection (NF1-TED) Study Page — https://www.nfresearch-childrens.org/